CLINICAL TRIAL: NCT02038894
Title: Comparison Of Different Anesthetic Techniques In Children Undergoing Esophagogastroduodenoscopies
Brief Title: Comparing Anesthetic Techniques in Children Having Esophagogastroduodenoscopies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2009-0100
Record Dates: First submitted 2013-05-01; First posted 2014-01-17 (Estimated); Results first posted 2020-09-24 (Actual); Last update posted 2020-09-24 (Actual); Status verified 2020-09

CONDITIONS: Eosinophilic Esophagitis
Keywords: Anesthetic; Pediatric; Esophagogastroduodenoscopies; Eosinophilic esophagitis; Gastroesophageal reflux disease (GERD); Abdominal Pain; Vomiting; Sevofluorane; Propofol; Nasal cannula; Intubation; Endotracheal tube
MeSH Terms: conditions — Eosinophilic Esophagitis; Gastroesophageal Reflux; Abdominal Pain; Vomiting | interventions — Sevoflurane; Propofol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Intubated with Sevoflurane (IS) (Active Comparator): Anesthetic technique during (EGD)
  Interventions: Drug: Intubated with Sevoflurane (IS)
- Intubated with Propofol (IP) (Active Comparator): Anesthetic technique during (EGD)
  Interventions: Drug: Intubated with Propofol (IP)
- Native Airway - no intubation (Active Comparator): Anesthetic technique during (EGD)
  Interventions: Drug: Zofran - no intubation; Drug: Propofol

INTERVENTIONS:
Drug: Intubated with Sevoflurane (IS) — Anesthesia will be maintained with sevoflurane 3% in oxygen at 2 L/min. The endoscopist will begin the procedure. The sevoflurane inspired concentration will be adjusted between 1 to 2 times the minimum alveolar concentration (MAC) by the attending anesthesiologist to maintain an appropriate level of anesthesia.
  Arms: Intubated with Sevoflurane (IS)
Drug: Intubated with Propofol (IP) — Anesthetic maintenance will be with 2 L/min flow of oxygen through the endotracheal tube and a continuous propofol infusion at a rate of 250 mcg/kg/min. A maximum of two bolus doses of propofol 0.5 to 1 mg/kg and an increase in the continuous infusion to 300 mcg/kg/min may be given at the discretion of the anesthetist if necessary to provide adequate anesthesia.
  Arms: Intubated with Propofol (IP)
Drug: Zofran - no intubation — A nasal cannula will be placed with oxygen administered at a rate of 3 L/min, and a bite block will be inserted. Zofran will be administered. Anesthesia will be maintained with a continuous propofol infusion at a rate of 250 mcg/kg/min. A maximum of two bolus doses of propofol 0.5 to 1 mg/kg, and an increase of the continuous infusion to 300 mcg/kg/min may be given at the discretion of the anesthetist.
  Arms: Native Airway - no intubation
Drug: Propofol
  Arms: Native Airway - no intubation

SUMMARY:
The purpose of this research study is to compare the safety and effectiveness of three commonly used techniques for delivering anesthesia during a procedure known as esophagogastroduodenoscopy.

DETAILED DESCRIPTION:
Different anesthetic techniques are currently in use at Cincinnati Children's Hospital Medical Center (CCHMC) for delivering anesthesia during an esophagogastroduodenoscopy (EGD). Because there is a lack of evidence to delineate the best techniques, pediatric anesthesiologists select the technique based on clinical preference and experience. One anesthetic technique involves the use of general anesthesia with the placement of an endotracheal tube, and maintenance with an inhalation agent, such as sevoflurane (IS). These patients may be extubated under deep anesthesia in the operating room, and allowed to awaken in the post anesthesia care unit. A similar technique involves the placement of an endotracheal tube, and anesthetic maintenance with a continuous infusion of propofol (IP). These patients are also extubated under deep anesthesia in the operating room, and allowed to awaken in the postoperative care unit. The third technique does not use an endotracheal tube and anesthetic maintenance occurs with continuous infusion of propofol with the patient breathing oxygen through their natural airway (NA). Our objective in this study is to compare outcomes between these three established anesthetic techniques.

Children in the study will be recruited from Cincinnati Children's Hospital Medical Center Operating Room Schedule. They will be cared for in the Operating Rooms and Post Anesthesia Care Unit.

ELIGIBILITY:
Inclusion Criteria:

* Patient presenting as out-patients, scheduled to receive an anesthetic for a diagnostic EGD
* Patient must be a candidate for any of the three anesthetic techniques. This decision will be made by a staff member of the Department of Anesthesiology, who is not a member of the study team and will be responsible for obtaining consent for anesthesia
* Patient must be between ages 1 and 12 years (inclusive)
* Patient must be American Society of Anesthesiology (ASA) class I or II;
* Eosinophilic esophagitis (EE) patients classified as an ASA III status for their EE diagnosis only
* Patient must have fasted according to CCHMC policy
* Patient's legally authorized representative has given written informed consent to participate in the study and, when appropriate, the subject has given assent to participate

Exclusion Criteria:

* Patients less than a year old and greater than 12 years old
* Patients undergoing therapeutic upper endoscopy
* Patients with an ASA physical status III or greater (other than EE patients)
* Patients with history of allergy to propofol, any other drug in the protocol, or eggs (exclusive of egg allergies identified only by skin testing or manifested only by gastrointestinal symptoms)
* Patients with personal or family history of malignant hyperthermia
* Obese patients (Body mass index more than 95th percentile for age)
* Patients with significant airway abnormalities (e.g., trisomy 21, craniofacial syndromes, sub-glottic stenosis, tracheomalacia, tracheostomy)
* Patients with history of obstructive sleep apnea
* Patient receiving sedative premedication
* Patient previously treated under this protocol
* Patients with symptoms of an active upper respiratory infection
* Patients with history of coagulopathy
* Patients with esophageal varices or gastrointestinal bleeding

Ages: 1 Year to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 179 (Actual)
Dates: Start 2009-12; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mario Patino, MD, Principal Investigator — Cincinati Children's Hospital Medical Center
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

REFERENCES:
- [Background] Hoffmann CO, Samuels PJ, Beckman E, Hein EA, Shackleford TM, Overbey E, Berlin RE, Wang Y, Nick TG, Gunter JB. Insufflation vs intubation during esophagogastroduodenoscopy in children. Paediatr Anaesth. 2010 Sep;20(9):821-30. doi: 10.1111/j.1460-9592.2010.03357.x. PMID 20716074
- [Background] Brown RH, Wagner EM. Mechanisms of bronchoprotection by anesthetic induction agents: propofol versus ketamine. Anesthesiology. 1999 Mar;90(3):822-8. doi: 10.1097/00000542-199903000-00025. PMID 10078684
- [Background] Oberer C, von Ungern-Sternberg BS, Frei FJ, Erb TO. Respiratory reflex responses of the larynx differ between sevoflurane and propofol in pediatric patients. Anesthesiology. 2005 Dec;103(6):1142-8. doi: 10.1097/00000542-200512000-00007. PMID 16306725
- [Background] Schwartz DA, Connelly NR, Theroux CA, Gibson CS, Ostrom DN, Dunn SM, Hirsch BZ, Angelides AG. Gastric contents in children presenting for upper endoscopy. Anesth Analg. 1998 Oct;87(4):757-60. doi: 10.1097/00000539-199810000-00003. PMID 9768765
- [Background] Lightdale JR, Mahoney LB, Schwarz SM, Liacouras CA. Methods of sedation in pediatric endoscopy: a survey of NASPGHAN members. J Pediatr Gastroenterol Nutr. 2007 Oct;45(4):500-2. doi: 10.1097/MPG.0b013e3180691168. PMID 18030225
- [Background] Elitsur Y, Blankenship P, Lawrence Z. Propofol sedation for endoscopic procedures in children. Endoscopy. 2000 Oct;32(10):788-91. doi: 10.1055/s-2000-7713. PMID 11068839
- [Background] Cravero JP, Blike GT, Beach M, Gallagher SM, Hertzog JH, Havidich JE, Gelman B; Pediatric Sedation Research Consortium. Incidence and nature of adverse events during pediatric sedation/anesthesia for procedures outside the operating room: report from the Pediatric Sedation Research Consortium. Pediatrics. 2006 Sep;118(3):1087-96. doi: 10.1542/peds.2006-0313. PMID 16951002
- [Background] Tosun Z, Aksu R, Guler G, Esmaoglu A, Akin A, Aslan D, Boyaci A. Propofol-ketamine vs propofol-fentanyl for sedation during pediatric upper gastrointestinal endoscopy. Paediatr Anaesth. 2007 Oct;17(10):983-8. doi: 10.1111/j.1460-9592.2007.02206.x. PMID 17767636
- [Background] Thakkar K, El-Serag HB, Mattek N, Gilger MA. Complications of pediatric EGD: a 4-year experience in PEDS-CORI. Gastrointest Endosc. 2007 Feb;65(2):213-21. doi: 10.1016/j.gie.2006.03.015. PMID 17258979
- [Background] Kaddu R, Bhattacharya D, Metriyakool K, Thomas R, Tolia V. Propofol compared with general anesthesia for pediatric GI endoscopy: is propofol better? Gastrointest Endosc. 2002 Jan;55(1):27-32. doi: 10.1067/mge.2002.120386. PMID 11756910
- [Background] U.S Food and Drug Administration. Med Watch. The FDA Safety Information and AdverseReportingProgram.Availableat:http://www.fda.gov/medWatch/report/DESK/advevnt.htm
- [Result] Patino M, Glynn S, Soberano M, Putnam P, Hossain MM, Hoffmann C, Samuels P, Kibelbek MJ, Gunter J. Comparison of different anesthesia techniques during esophagogastroduedenoscopy in children: a randomized trial. Paediatr Anaesth. 2015 Oct;25(10):1013-9. doi: 10.1111/pan.12717. Epub 2015 Jul 17. PMID 26184697

RESULTS

PARTICIPANT FLOW:
Groups:
- Native Airway - no Intubation: Anesthetic technique during (EGD)
  Zofran - no intubation: A nasal cannula will be placed with oxygen administered at a rate of 3 L/min, and a bite block will be inserted. Zofran will be administered. Anesthesia will be maintained with a continuous propofol infusion at a rate of 250 mcg/kg/min. A maximum of two bolus doses of propofol 0.5 to 1 mg/kg, and an increase of the continuous infusion to 300 mcg/kg/min may be given at the discretion of the anesthetist.
  Propofol
Period: Overall Study
Arm/Group | Intubated With Sevoflurane (IS) | Intubated With Propofol (IP) | Native Airway - no Intubation
Started | 60 | 58 | 61
Completed | 60 | 58 | 61
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intubated With Sevoflurane (IS) | Intubated With Propofol (IP) | Native Airway - no Intubation | Total
Number analyzed (Participants) | 60 | 58 | 61 | 179
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 8 [4 to 10] | 6 [4 to 9] | 7 [4 to 10] | 7 [4 to 10]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 25 | 26 | 78
  Male | 33 | 33 | 35 | 101
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American | 4 | 2 | 2 | 8
  Asian | 1 | 1 | 1 | 3
  Caucasian | 55 | 52 | 51 | 158
  Other | 0 | 2 | 6 | 8
  Unknown | 0 | 1 | 1 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 60 | 58 | 61 | 179
Weight [Median (Inter-Quartile Range); unit: kg] | 25 [15.9 to 35.8] | 22.7 [17.8 to 31.8] | 22.5 [16.5 to 37.7] | 24.3 [16.4 to 35.3]
BMI [Median (Inter-Quartile Range); unit: kg/m^2] | 16 [14.9 to 17.9] | 16.1 [14.8 to 17.4] | 16.6 [15.3 to 18.4] | 16.4 [15 to 17.9]
BMI Percent [Median (Inter-Quartile Range); unit: percentile] | 46 [21.6 to 78.2] | 57.1 [24.6 to 76.9] | 67 [39.9 to 83.7] | 56.8 [25.3 to 81.7]
American Society of Anesthesiologists - ASA Physical Status (Patient's health condition) [Count of Participants; unit: Participants]
  ASA 1 (Normal healthy subject) | 13 | 15 | 10 | 38
  ASA 2 (Mild systemic disease) | 47 | 43 | 50 | 140
  Missing or Unknown | 0 | 0 | 1 | 1
Diagnosis [Count of Participants; unit: Participants]
  Abdominal Pain | 15 | 20 | 15 | 50
  Chronic Diarrhea | 3 | 3 | 1 | 7
  Diarrhea | 1 | 1 | 0 | 2
  Dysphagia | 4 | 3 | 0 | 7
  Eosinophilic esophagitis | 18 | 10 | 24 | 52
  Failure to Thrive | 5 | 3 | 5 | 13
  Feeding Difficulties | 2 | 1 | 0 | 3
  GERD | 6 | 5 | 8 | 19
  Nausea/Vomit | 4 | 9 | 7 | 20
  Rumination Syndrome | 0 | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Respiratory Complications
Description: An important outcome in the anesthetic management of these patients is to maintain a balance between a safe technique with a minimal incidence of respiratory complications, and a technique that facilitates rapid turnover of the gastrointestinal suite. A chi-square test, or Fisher's exact test will measure differences among the three anesthetic groups. Different anesthetic techniques are currently in use at Cincinnati Children's Hospital Medical Center (CCHMC). Because there is a lack of evidence to delineate the best techniques, pediatric anesthesiologists select the technique based on clinical preference and experience.
Time Frame: Admission for surgery through recovery period, approximately 3 hours
Measure: Count of Participants; unit: Participants
Groups:
- IS and IP: Grouping the intubated with sevoflurane group (IS) with the intubated with propofol group (IP) since the airway management is the same for both groups (endotracheal intubation) Table 2
- IP and NA: Grouping the intubated propofol group (IP) with the native airway group (NA) since they received the same medication during the procedure (propofol). Table 2
Arm/Group | Intubated With Sevoflurane (IS) | Intubated With Propofol (IP) | Native Airway - no Intubation | IS and IP | IP and NA
Number analyzed (Participants) | 60 | 58 | 61 | 118 | 119
Participants
  SPO2 < 95% | 0 | 0 | 15 | 0 | 15
  SPO2 < 85% | 0 | 0 | 9 | 0 | 8
  Apnea | 0 | 1 | 5 | 1 | 5
  Inadequate Anesthesia | 1 | 4 | 9 | 5 | 13
  All Respiratory Events | 2 | 5 | 28 | 7 | 32
Statistical Analysis 1: Comparison: Native Airway - no Intubation vs IS and IP; Test type: Non-Inferiority — A previous study for evaluating respiratory complications with intubated and insufflated techniques found a difference in the incidence of respiratory complications of 9.1%, a power analysis was determined. 200 subjects per group was estimated provide 82% power to detect a difference. We elected to do an interim analysis when 60 children per group were recruited because of a clinical impression that one of the techniques had a grossly divergent incidence of respiratory complications; p < 0.0001, Mean equality test — Threshold for significance <0.05 Comparing SPO2 <95%; Odds Ratio (OR) = 0, 95% CI 2-sided [0 to 0.14]
Statistical Analysis 2: Comparison: Intubated With Sevoflurane (IS) vs Intubated With Propofol (IP) vs Native Airway - no Intubation vs IS and IP vs IP and NA; Test type: Non-Inferiority — A previous study found an incidence of respiratory complications of 9.1%. 200 subjects per group was estimated provide 82% power to detect a difference when conducting a two- sided test at a significance level of a = 0.05.We did an interim analysis when 60 children per group were recruited because of a clinical impression that one of the techniques had a grossly divergent incidence of respiratory complications. Based on the results of that interim analysis, recruitment was discontinued; p = 0.0001, Mean equality test — p<0.05. Sp02<85%; Odds Ratio (OR) = 0, 95% CI 2-sided [0 to 0.27] — Odds ratios were calculated to the respiratory complications comparing the different groups and by regrouping by the differences in airway management (IS + IP vs NA) and by the medication used for anesthesia maintenance (IS vs IP + NA)

2. Secondary Outcome: Peri-operative Times Between Three Different Anesthetic Techniques
Description: Time measurements are used to evaluate the efficiency of the different techniques. We will compare the times spent in the operating room and the postoperative unit for each technique.
Time Frame: Admission for surgery through recovery period, approximately 3 hours
Measure: Mean (Standard Deviation); unit: Minutes
Groups:
- IS and IP: Grouped together by the same airway management during anesthesia (Endotracheal intubation). Table 2
- IP and NA: Grouped together by the same medication use for anesthesia maintenance (propofol). Table 2
Arm/Group | Intubated With Sevoflurane (IS) | Intubated With Propofol (IP) | Native Airway - no Intubation | IS and IP | IP and NA
Number analyzed (Participants) | 60 | 58 | 61 | 118 | 119
Minutes
  OR Time | 24.03 (6.00) | 24.19 (7.54) | 23.05 (7.97) | 24.11 (6.77) | 23.61 (7.75)
  Anesthesia Preparation Time | 10.86 (2.53) | 10.70 (2.70) | 10.35 (3.35) | 10.78 (2.60) | 10.53 (3.03)
  Procedural Time | 9.07 (4.78) | 9.23 (5.46) | 8.33 (4.18) | 9.15 (5.11) | 8.78 (4.86)
  PACU efficiency time | 49.50 (14.31) | 53.49 (12.68) | 54.42 (22.59) | 51.48 (13.61) | 53.96 (18.24)
  Total Perioperative Time | 75.34 (15.40) | 79.61 (14.45) | 79.37 (25.17) | 77.46 (15.03) | 79.49 (20.43)
Statistical Analysis 1: Comparison: Intubated With Sevoflurane (IS) vs Intubated With Propofol (IP) vs Native Airway - no Intubation vs IS and IP vs IP and NA; Total OR Time; Test type: Non-Inferiority — No previous data was available to calculate a power calculation for the secondary outcome; p = 0.901, Mean equality test — Threshold of Significance

ADVERSE EVENTS:
Arm/Group | Intubated With Sevoflurane (IS) | Intubated With Propofol (IP) | Native Airway - no Intubation
Serious Adverse Events (participants affected / at risk) | 0/60 | 1/58 | 14/61
Other Adverse Events (participants affected / at risk) | 1/60 | 4/58 | 24/61
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intubated With Sevoflurane (IS) (N=60) | Intubated With Propofol (IP) (N=58) | Native Airway - no Intubation (N=61)
Severe desaturation: SpO2 < 85% (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 9 (9) — A recorded SpO2 < 85% during the anesthesia
Apnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 5 (5)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intubated With Sevoflurane (IS) (N=60) | Intubated With Propofol (IP) (N=58) | Native Airway - no Intubation (N=61)
Minor desaturation < 95% (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 15 (15)
Inadequate anesthesia (Surgical and medical procedures) | 1 (1) | 4 (4) | 9 (9)

LIMITATIONS AND CAVEATS:
prior to conclusion. THis is optional

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No